CLINICAL TRIAL: NCT03931798
Title: The Visual Scanning Test: a Neuropsychological Tool to Assess Extrapersonal Visual Unilateral Spatial Neglect
Acronym: VST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: Rehabilitation Istitute Santa Maria Bambina (Unknown); Clinical Center Agoretis (Unknown)
Responsible Party: Principal Investigator, Francesca Cecchi, Dr, Fondazione Don Carlo Gnocchi Onlus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRCCSdongnocchi
Record Dates: First submitted 2019-04-26; First posted 2019-04-30 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Spatial Neglect
Keywords: Unilateral spatial neglect; Extrapersonal space; Neuropsychology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Healthy participants were administered the Visual Scanning Test
  Interventions: Diagnostic Test: Visual Scanning Test

INTERVENTIONS:
Diagnostic Test: Visual Scanning Test — The Visual Scanning Test (VST) involved a visual search for a target between similar visual distractors, projected in the far space, so as to simulate the search within a visual field. It is overall composed by four trials, each trial contained 20 cases and made up by 20 stimuli. On about the 80% of cases, the test provided the presence of target in the left, center or in right hemispace. In the remaining 20% of cases, the test provided the presence of a catch trial (absence of the target), to assess the presence of frontal disturbances or malingering. The test is constructed according to an increasing attentional load for the target on the left-hemispace. Participants, sitting in front a blank wall, were required to actively and free explore the projected visual field to search for the visual target, naming its identification (saying YES or NO). During the task, the examiner annotated the reaction times and the errors.

SUMMARY:
Presentation and standardization on a normative sample of a new neuropsychological tool to provide a quantitative assessment of visual unilateral spatial neglect in the extrapersonal portion of space.

DETAILED DESCRIPTION:
Unilateral spatial neglect (USN) represents one of the most frequent and disabling neuropsychological consequences of acute brain damage. Patients with USN show an impaired ability to perceive sensory events and to perform actions in the contralesional side of the space, in absence of a lower-level sensory or motor deficit. Several studies found that controlesional USN is more frequent and more severe in right than left parietal damage and due to its prominent impairment, USN has broadly been studied in the visual modality (VUSN). VUSN can affect patient's own contralesional body (personal neglect), into the near space within reaching distance (peripersonal) or space beyond reaching distance (far extrapersonal space). Those portions of space may dissociate and patient may show extrapersonal VUSN without alterations on the other portions of space (i.e. personal and peripersonal). Traditional paper-and-pencil neuropsychological tests are useful and widely used to evaluate VUSN, even if several of them can provide an assessment of peripersonal VUSN. In fact, this portion of space can be assessed through line bisection, cancellation, or copy tasks which are normally completed within reaching distance. Instead, personal and extrapersonal neglect are less easily evaluated: this lack of assessment tools may lead to lower detection rates for USN in patients in clinical setting and lead to relevant clinical implications. Finally, paper-and-pencil tests can detect only a moderate or even severe deficit due to VUSN but not a mild impairment and they are not informative about patients' disability in natural setting. According to this limitations of traditional paper-and-pencil tests, several studies have shown that computerized reaction time tasks are more sensitive in the detection of lateralized spatial attention deficits in patients with mild or remitted VUSN. The primary aim of this study was to present and standardize a new neuropsychological tool to provide a quantitative assessment of VUSN in the extrapersonal portion of space.

The Visual Scanning Test (VST) involved a visual search for a target between similar visual distractors, projected in the far space, so as to simulate the search within a visual field. It is overall composed by four trials, each trial contained 20 cases and made up by 20 stimuli. On about the 80% of cases, the test provided the presence of target in the left, center or in right hemispace. In the remaining 20% of cases, the test provided the presence of a catch trial (absence of the target), to assess the presence of frontal disturbances or malingering. The test is constructed according to an increasing attentional load for the target on the left-hemispace. Participants, sitting in front a blank wall, were required to actively and free explore the projected visual field to search for the visual target, naming its identification (saying YES or NO). During the task, the examiner annotated the reaction times and the errors. From these data it was possible to get some informative indexes regarding the reaction times, the accuracy and the implicit learning of the progressive shift to the left of the target and the possible presence of asymmetry in the visual exploration.

ELIGIBILITY:
Inclusion Criteria:

- healthy subjects of full age.

Exclusion Criteria:

* past or present neurological diseases;
* past or present psychiatric diseases;
* presence of visual disturbances.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2015-11-02 (Actual); Primary Completion 2017-01-15 (Actual); Study Completion 2018-01-09 (Actual)

PRIMARY OUTCOMES:
Scores of clinical indexes due to the accuracy and the reaction times | Clinical indexes were obtained after completing th edata collecyion, which lasted two years
  From the obtained data it was possible to get some informative indexes regarding the reaction times, the accuracy and the implicit learning of the progressive shift to the left of the target and the possible presence of asymmetry in the visual exploration.

IPD SHARING:
Plan to Share IPD: No
We didn't plan to share these data

REFERENCES:
- [Background] Priftis K, Passarini L, Pilosio C, Meneghello F, Pitteri M. Visual Scanning Training, Limb Activation Treatment, and Prism Adaptation for Rehabilitating Left Neglect: Who is the Winner? Front Hum Neurosci. 2013 Jul 8;7:360. doi: 10.3389/fnhum.2013.00360. eCollection 2013. PMID 23847520
- [Background] Vallar G, Calzolari E. Unilateral spatial neglect after posterior parietal damage. Handb Clin Neurol. 2018;151:287-312. doi: 10.1016/B978-0-444-63622-5.00014-0. PMID 29519463
- [Background] Vallar, G., & Bolognini, N. (2014). Unilateral spatial neglect. In A. C. Nobre & S. Kastner (Eds.), Oxford library of psychology. The Oxford handbook of attention (pp. 972-1027). New York, NY, US: Oxford University Press..
- [Background] Bisiach E, Vallar G, Perani D, Papagno C, Berti A. Unawareness of disease following lesions of the right hemisphere: anosognosia for hemiplegia and anosognosia for hemianopia. Neuropsychologia. 1986;24(4):471-82. doi: 10.1016/0028-3932(86)90092-8. PMID 3774133
- [Background] Ten Brink AF, Verwer JH, Biesbroek JM, Visser-Meily JMA, Nijboer TCW. Differences between left- and right-sided neglect revisited: A large cohort study across multiple domains. J Clin Exp Neuropsychol. 2017 Sep;39(7):707-723. doi: 10.1080/13803395.2016.1262333. Epub 2016 Dec 12. PMID 27951747
- [Background] Ten Brink AF, Biesbroek JM, Oort Q, Visser-Meily JMA, Nijboer TCW. Peripersonal and extrapersonal visuospatial neglect in different frames of reference: A brain lesion-symptom mapping study. Behav Brain Res. 2019 Jan 1;356:504-515. doi: 10.1016/j.bbr.2018.06.010. Epub 2018 Jun 22. PMID 29940260
- [Background] Bowen A, McKenna K, Tallis RC. Reasons for variability in the reported rate of occurrence of unilateral spatial neglect after stroke. Stroke. 1999 Jun;30(6):1196-202. doi: 10.1161/01.str.30.6.1196. PMID 10356099
- [Background] Denes G, Semenza C, Stoppa E, Lis A. Unilateral spatial neglect and recovery from hemiplegia: a follow-up study. Brain. 1982 Sep;105 (Pt 3):543-52. doi: 10.1093/brain/105.3.543. PMID 7104665
- [Background] Machner B, Konemund I, von der Gablentz J, Bays PM, Sprenger A. The ipsilesional attention bias in right-hemisphere stroke patients as revealed by a realistic visual search task: Neuroanatomical correlates and functional relevance. Neuropsychology. 2018 Oct;32(7):850-865. doi: 10.1037/neu0000493. PMID 30321035
- [Background] Gainotti G. The role of automatic orienting of attention towards ipsilesional stimuli in non-visual (tactile and auditory) neglect: a critical review. Cortex. 2010 Feb;46(2):150-60. doi: 10.1016/j.cortex.2009.04.006. Epub 2009 May 14. PMID 19501350
- [Background] Appelros P, Nydevik I, Karlsson GM, Thorwalls A, Seiger A. Assessing unilateral neglect: shortcomings of standard test methods. Disabil Rehabil. 2003 May 6;25(9):473-9. doi: 10.1080/0963828031000071714. PMID 12745942
- [Background] Buxbaum LJ, Ferraro MK, Veramonti T, Farne A, Whyte J, Ladavas E, Frassinetti F, Coslett HB. Hemispatial neglect: Subtypes, neuroanatomy, and disability. Neurology. 2004 Mar 9;62(5):749-56. doi: 10.1212/01.wnl.0000113730.73031.f4. PMID 15007125
- [Background] Danckert J, Ferber S. Revisiting unilateral neglect. Neuropsychologia. 2006;44(6):987-1006. doi: 10.1016/j.neuropsychologia.2005.09.004. Epub 2005 Nov 21. PMID 16300805
- [Background] Berti A, Smania N, Rabuffetti M, Ferrarin M, Spinazzola L, D'Amico A, Ongaro E, Allport A. Coding of far and near space during walking in neglect patients. Neuropsychology. 2002 Jul;16(3):390-9. doi: 10.1037//0894-4105.16.3.390. PMID 12146686
- [Background] Lindell AB, Jalas MJ, Tenovuo O, Brunila T, Voeten MJ, Hamalainen H. Clinical assessment of hemispatial neglect: evaluation of different measures and dimensions. Clin Neuropsychol. 2007 May;21(3):479-97. doi: 10.1080/13854040600630061. PMID 17455032
- [Background] Pedroli E, Serino S, Cipresso P, Pallavicini F, Riva G. Assessment and rehabilitation of neglect using virtual reality: a systematic review. Front Behav Neurosci. 2015 Aug 25;9:226. doi: 10.3389/fnbeh.2015.00226. eCollection 2015. PMID 26379519
- [Background] Parton A, Malhotra P, Husain M. Hemispatial neglect. J Neurol Neurosurg Psychiatry. 2004 Jan;75(1):13-21. PMID 14707298
- [Background] Coslett HB. Apraxia, Neglect, and Agnosia. Continuum (Minneap Minn). 2018 Jun;24(3, BEHAVIORAL NEUROLOGY AND PSYCHIATRY):768-782. doi: 10.1212/CON.0000000000000606. PMID 29851877
- [Background] Butler BC, Eskes GA, Vandorpe RA. Gradients of detection in neglect: comparison of peripersonal and extrapersonal space. Neuropsychologia. 2004;42(3):346-58. doi: 10.1016/j.neuropsychologia.2003.08.008. PMID 14670573
- [Background] Cipresso P, Pedroli E, Serino S, Semonella M, Tuena C, Colombo D, Pallavicini F, Riva G. Assessment of Unilateral Spatial Neglect Using a Free Mobile Application for Italian Clinicians. Front Psychol. 2018 Nov 22;9:2241. doi: 10.3389/fpsyg.2018.02241. eCollection 2018. PMID 30524341
- [Background] Cocchini, G., Beschin, N., &Jehkonen, M. (2001). The Fluff Test: A simple task to assess body representation neglect. Neuropsychological Rehabilitation, 11(1), 17-31.
- [Background] Azouvi P, Olivier S, de Montety G, Samuel C, Louis-Dreyfus A, Tesio L. Behavioral assessment of unilateral neglect: study of the psychometric properties of the Catherine Bergego Scale. Arch Phys Med Rehabil. 2003 Jan;84(1):51-7. doi: 10.1053/apmr.2003.50062. PMID 12589620
- [Background] Rengachary J, d'Avossa G, Sapir A, Shulman GL, Corbetta M. Is the posner reaction time test more accurate than clinical tests in detecting left neglect in acute and chronic stroke? Arch Phys Med Rehabil. 2009 Dec;90(12):2081-8. doi: 10.1016/j.apmr.2009.07.014. PMID 19969172
- [Background] Cunningham LJ, O'Rourke K, Finlay C, Gallagher M. A preliminary investigation into the psychometric properties of the Dublin Extrapersonal Neglect Assessment (DENA): A novel screening tool for extrapersonal neglect. Neuropsychol Rehabil. 2017 Apr;27(3):349-368. doi: 10.1080/09602011.2015.1084334. Epub 2015 Sep 30. PMID 26421958
- [Background] Bonato M. Neglect and extinction depend greatly on task demands: a review. Front Hum Neurosci. 2012 Jul 17;6:195. doi: 10.3389/fnhum.2012.00195. eCollection 2012. PMID 22822394
- [Background] Barrett AM, Buxbaum LJ, Coslett HB, Edwards E, Heilman KM, Hillis AE, Milberg WP, Robertson IH. Cognitive rehabilitation interventions for neglect and related disorders: moving from bench to bedside in stroke patients. J Cogn Neurosci. 2006 Jul;18(7):1223-36. doi: 10.1162/jocn.2006.18.7.1223. PMID 16839294
- [Background] Hasegawa C, Hirono N, Yamadori A. Discrepancy in unilateral spatial neglect between daily living and neuropsychological test situations: a single case study. Neurocase. 2011 Dec;17(6):518-26. doi: 10.1080/13554794.2010.547506. Epub 2011 Jun 27. PMID 21707261
- [Background] Bonato M, Priftis K, Marenzi R, Umilta C, Zorzi M. Deficits of contralesional awareness: a case study on what paper-and-pencil tests neglect. Neuropsychology. 2012 Jan;26(1):20-36. doi: 10.1037/a0025306. Epub 2011 Sep 5. PMID 21895377
- [Background] Bonato M, Deouell LY. Hemispatial neglect: computer-based testing allows more sensitive quantification of attentional disorders and recovery and might lead to better evaluation of rehabilitation. Front Hum Neurosci. 2013 May 1;7:162. doi: 10.3389/fnhum.2013.00162. eCollection 2013. No abstract available. PMID 23641207
- [Background] Priftis K, Bonato M, Zorzi M, Umilta C. Spatial and non-spatial aspects of neglect. Front Hum Neurosci. 2013 Feb 5;7:25. doi: 10.3389/fnhum.2013.00025. eCollection 2013. No abstract available. PMID 23386825
- [Background] Kerkhoff G, Schenk T. Rehabilitation of neglect: an update. Neuropsychologia. 2012 May;50(6):1072-9. doi: 10.1016/j.neuropsychologia.2012.01.024. Epub 2012 Jan 28. PMID 22306520
- [Background] Capitani, E. (1997). Normative data and neuropsychological assessment. Common problems in clinical practice and research. Neuropsychological Rehabilitation, 7(4), 295-310.
- [Background] Capitani E, Laiacona M. Composite neuropsychological batteries and demographic correction: standardization based on equivalent scores, with a review of published data. The Italian Group for the Neuropsychological Study of Ageing. J Clin Exp Neuropsychol. 1997 Dec;19(6):795-809. doi: 10.1080/01688639708403761. PMID 9524875
- [Background] Wilks, S. S. (1941). Determination of sample sizes for setting tolerance limits. The Annals of Mathematical Statistics, 12(1), 91-96.
- [Background] Capitani E, Laiacona M. Outer and inner tolerance limits: their usefulness for the construction of norms and the standardization of neuropsychological tests. Clin Neuropsychol. 2017 Aug-Oct;31(6-7):1219-1230. doi: 10.1080/13854046.2017.1334830. Epub 2017 Jun 9. PMID 28598726
- [Background] Bartolomeo P, Chokron S. Left unilateral neglect or right hyperattention? Neurology. 1999 Dec 10;53(9):2023-7. doi: 10.1212/wnl.53.9.2023. PMID 10599775
- [Background] Bartolomeo, P. (2014). The attention systems of the human brain. In Attention Disorders After Right Brain Damage (pp. 1-19). Springer, London.
- [Background] Bourgeois A, Chica AB, Migliaccio R, Thiebaut de Schotten M, Bartolomeo P. Cortical control of inhibition of return: evidence from patients with inferior parietal damage and visual neglect. Neuropsychologia. 2012 Apr;50(5):800-9. doi: 10.1016/j.neuropsychologia.2012.01.014. Epub 2012 Jan 20. PMID 22285795
- [Result] Posner MI, Walker JA, Friedrich FJ, Rafal RD. Effects of parietal injury on covert orienting of attention. J Neurosci. 1984 Jul;4(7):1863-74. doi: 10.1523/JNEUROSCI.04-07-01863.1984. PMID 6737043
- [Result] Lupianez J, Klein RM, Bartolomeo P. Inhibition of return: Twenty years after. Cogn Neuropsychol. 2006 Oct 1;23(7):1003-14. doi: 10.1080/02643290600588095. PMID 21049364
- [Result] Hartmann M, Sommer NR, Diana L, Muri RM, Eberhard-Moscicka AK. Further to the right: Viewing distance modulates attentional asymmetries ('pseudoneglect') during visual exploration. Brain Cogn. 2019 Feb;129:40-48. doi: 10.1016/j.bandc.2018.11.008. Epub 2018 Nov 22. PMID 30471991
- [Result] Gamberini L, Seraglia B, Priftis K. Processing of peripersonal and extrapersonal space using tools: evidence from visual line bisection in real and virtual environments. Neuropsychologia. 2008 Apr;46(5):1298-304. doi: 10.1016/j.neuropsychologia.2007.12.016. Epub 2007 Dec 27. PMID 18242649
- [Result] Bjoertomt O, Cowey A, Walsh V. Spatial neglect in near and far space investigated by repetitive transcranial magnetic stimulation. Brain. 2002 Sep;125(Pt 9):2012-22. doi: 10.1093/brain/awf211. PMID 12183347
- [Result] Heilman KM, Van Den Abell T. Right hemisphere dominance for attention: the mechanism underlying hemispheric asymmetries of inattention (neglect). Neurology. 1980 Mar;30(3):327-30. doi: 10.1212/wnl.30.3.327. PMID 7189037
- [Result] Mesulam MM. Spatial attention and neglect: parietal, frontal and cingulate contributions to the mental representation and attentional targeting of salient extrapersonal events. Philos Trans R Soc Lond B Biol Sci. 1999 Jul 29;354(1387):1325-46. doi: 10.1098/rstb.1999.0482. PMID 10466154
- [Derived] Borsotti M, Mosca IE, Di Lauro F, Pancani S, Bracali C, Dore T, Macchi C, Cecchi F; IRCCS Don Gnocchi Stroke Group. The Visual Scanning Test: a newly developed neuropsychological tool to assess and target rehabilitation of extrapersonal visual unilateral spatial neglect. Neurol Sci. 2020 May;41(5):1145-1152. doi: 10.1007/s10072-019-04218-2. Epub 2020 Jan 2. PMID 31897939

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-09): https://cdn.clinicaltrials.gov/large-docs/98/NCT03931798/Prot_SAP_000.pdf